CLINICAL TRIAL: NCT05630638
Title: Doravirine Dose Optimisation in Pregnancy
Acronym: DoraDO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool School of Tropical Medicine (Other); Desmond Tutu Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UoL001707
Record Dates: First submitted 2022-09-14; First posted 2022-11-29 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: HIV
Keywords: Pregnancy
MeSH Terms: interventions — doravirine; dolutegravir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delstrigo (Experimental): doravirine/lamivudine/tenofovir disoproxil 100 mg/ 300 mg/ 245 mg film coated tablets, dosed 1 tablet once daily for the duration of the study
  Interventions: Drug: Doravirine
- Standard of care (Active Comparator): dolutegravir/lamivudine/tenofovir disoproxil 50 mg/300 mg/245 mg film coated tablets, dosed 1 tablet once daily for the duration of the study
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Doravirine — Fixed dose combination of doravirine, lamivudine and tenofovir disoproxil
  Other Names: Delstrigo
  Arms: Delstrigo
Drug: Dolutegravir — Fixed dose combination of dolutegravir, lamivudine and tenofovir disoproxil
  Other Names: TLD
  Arms: Standard of care

SUMMARY:
A randomised, open label, controlled PK standard of care vs doravirine plus 2 nucleoside reverse transcriptase inhibitors backbone in pregnant women initiating combination antiretroviral therapy in the second trimester of pregnancy.

DETAILED DESCRIPTION:
Women diagnosed HIV positive in the second trimester of pregnancy in South Africa will be enrolled and randomised 1:1 to receive standard of care or doravirine plus 2 NRTI backbone. Participants will receive study treatment until delivery and up to 28 weeks postpartum, with a maximum total of 14 months of study treatment. Given the high prevalence of NNRTI resistance, alternative ARV treatment options are essential. Doravirine is licenced for the treatment of HIV-1 in adults in North America and Europe. Whilst the efficacy and safety of doravirine has been established in non-pregnant adults, there are no adequate human data available to establish whether DOR poses a risk to pregnancy outcomes. It is important to have data on the safety and pharmacokinetics of the drug during pregnancy and in particularly the third trimester of pregnancy in order to support its use. The hypothesis for this study is that pregnancy influences the pharmacokinetics of doravirine when initiated in the second trimester.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old
* Ability to give informed consent prior to participation
* Willing and able to comply with all study requirements
* HIV positive
* Pregnant (initiating cART ≥ 12 weeks and < 26 weeks gestation)
* Intention to breastfeed postpartum

Exclusion Criteria:

* Received any cART in preceding 6 months
* Chronic hepatitis B (HBV) infection with clinical evidence of transaminitis
* Elevations in serum levels of alanine aminotransferase (ALT) > 5 times the upper limit of normal (ULN) or ALT > 3xULN and bilirubin >2xULN (with > 35 % direct bilirubin)
* Previous documented failure of an NNRTI-containing cART regimen
* Previous history of hypersensitivity to any ARV
* Concomitant medication which are inducers of SoC and DOR metabolism (e.g. rifampicin, anti-epileptic agents, rifabutin, St John's Wort, mitotane, enzalutamide, lumacaftor). Contraindicated medications can be found on Liverpool Drug Interactions website (hiv-druginteractions.org)
* Participants with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption cannot take DOR as the tablet contains lactose monohydrate
* Clinical depression or clinical judgment suggests increased risk of suicidality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
AUC of doravirine in pregnant women | 24 to 28 weeks gestation, 32 to 36 weeks gestation, 6 weeks postpartum
  Pharmacokinetic parameters of doravirine in pregnancy - AUC
Cmax of doravirine in pregnant women | 24 to 28 weeks gestation, 32 to 36 weeks gestation, 6 weeks postpartum
  Pharmacokinetic parameters of doravirine in pregnancy - Cmax
Cmin of doravirine in pregnant women | 24 to 28 weeks gestation, 32 to 36 weeks gestation, 6 weeks postpartum
  Pharmacokinetic parameters of doravirine in pregnancy - Cmin
CL/F of doravirine in pregnant women | 24 to 28 weeks gestation, 32 to 36 weeks gestation, 6 weeks postpartum
  Pharmacokinetic parameters of doravirine in pregnancy - CL/F

SECONDARY OUTCOMES:
To assess the number of treatment related adverse events by DAIDS v2.1 | Until study completion, a maximum of 13 months
  Safety and tolerability of doravirine in mothers and neonates
To determine the concentration of doravirine in breastmilk, in breastfed infants, in genital tract, cord blood | 24 to 28 weeks gestation, 32 to 36 weeks gestation, 6 weeks postpartum
  Pharmacokinetics of doravirine in various compartments
To assess maternal viral load responses | Delivery and 6 months postpartum
  Viral load assessment
To determine infant transmissions in the first 6 months of life using HIV viral load | Delivery until 6 months postpartum
  Assessment of perinatal transmission using HIV viral load
To assess the prevalence or emergence of HIV drug resistance by determining HIV mutations | Until study completion, a maximum of 13 months
  Assessment of drug resistance tests

OTHER OUTCOMES:
Viral dynamics in the genital tract of mothers | Baseline and 32 to 36 weeks gestation
  Assessment of viral load in the genital tract
PK in the genital tract of mothers | Baseline and 32 to 36 weeks gestation
  Assessment of drug concentrations in the genital tract
PK of DOR in breastmilk, breastfed infants and in the genital tract | Delivery, 6 weeks postpartum and 24 weeks postpartum
  Assessment of drug concentrations in non-plasma compartments
Prevalence or emergence of HIV drug resistance by determining HIV mutations | Baseline to 24 weeks postpartum
  Assessment of drug resistance tests

CONTACTS AND LOCATIONS:
Overall Officials: Saye Khoo, Principal Investigator — University of Liverpool
Locations (1):
- Desmond Tutu Health Foundation, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The investigators will consider all reasonable requests by health-care providers, investigators, and researchers to provide anonymised data to address specific scientific or clinical objectives. The investigators are committed to reviewing requests from researchers for access to clinical trial protocols, de-identified patient-level clinical trial data, and study-level clinical trial data. Data will be assigned a DOI through deposition in the University of Liverpool Research Data Catalogue (rdm@liverpool.ac.uk) and shared under a Data Transfer agreement (or equivalent e.g. as part of a research collaboration agreement or confidentiality disclosure agreement).
Supporting Information: Study Protocol
Time Frame: After study analysis has completed and manuscript is published for at least 5 years afterwards.
Access Criteria: By reasonable request to the investigators.